CLINICAL TRIAL: NCT06629805
Title: Effect of Aureobasidium Pullulans Produced β-glucan and Regular Combined Exercise on Musculoskeletal Function and Biomarkers in Adults With Relative Sarcopenia: a Randomized Controlled Trial
Brief Title: β-glucan and Exercise on Musculoskeletal Function in Sarcopenic Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-2024-003
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aureobasidium pullulans produced β-glucan group (Experimental): This group takes Aureobasidium pullulans produced β-glucan for 12 weeks.
  Interventions: Dietary Supplement: Aureobasidium pullulans produced β-glucan
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aureobasidium pullulans produced β-glucan — Aureobasidium pullulans produced β-glucan 1,000 mg/day for 12 weeks
  Arms: Aureobasidium pullulans produced β-glucan group
Dietary Supplement: Placebo — Placebo 1,000 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Aureobasidium pullulans produced β-glucan and regular combined exercise on muscle strength, muscle mass, muscle function, and biomarkers in adults with relative sarcopenia for 12 weeks.

DETAILED DESCRIPTION:
A previous human study has indicated that Aureobasidium pullulans produced β-glucan may increase muscle mass and strength in the elderly. Therefore, the investigators will conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Aureobasidium pullulans produced β-glucan on muscle strength, muscle mass, and muscle function, expanding the target population to adults aged 50 and older with relative sarcopenia, the safety of the compound are also evaluated. The Investigators examine the peak torque/body weight at 60°/s knee extension, handgrip strength, skeletal muscle mass, physical performance, and metabolic parameters at baseline and 12 weeks of intervention. Eighty adults were administered either 1,000 mg of Aureobasidium pullulans produced β-glucan or a placebo each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* <110% of the standard lean body mass as measured using the body composition analyzer
* Body mass index (BMI) ranging from 18.5 to 30.0 kg/m2
* Grip strength of the frequently used hand is based on the following age-specific standards: Men in their 50s (less than 42 kg, women: less than 25.1 kg), Men in their 60s (less than 38.5 kg, women: less than 24.1 kg), Men 70 and older (less than 33.2 kg, women: less than 20.9 kg)
* Individuals with a Short Physical Performance Battery score of 9 or higher.

Exclusion Criteria:

* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* History of fracture during the previous year
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* History of serious cerebro-cardiovascular diseases or cancer such as angina or myocardial infarction within 6 months
* History of any central bone fracture within 1 year
* History of medication for psychiatric diseases such as severe depression, schizophrenia, and drug intoxication.
* Alcohol abuser
* Allergic reaction to Aureobasidium pullulans produced β-glucan
* Those who participated in other drug clinical trials within 1 month from the screening date.
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or plan to become pregnant during the clinical trial
* Those who are judged to be unsuitable by the PI for other reasons

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 12 weeks
  The peak torque at 60°/s knee extension (/kg), right, left and the peak torque at 60°/s knee flexion (/kg), right, left
TUG test | 12 weeks
  Timed Up & Go test

SECONDARY OUTCOMES:
Appendicular skeletal mass/(height x height) | 12 weeks
  Using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
Appendicular skeletal mass/weight x 100 | 12 weeks
  Using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
Skeletal Muscle Mass Index/(height x height) | 12 weeks
  Using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
Hand grip strength, both | 12 weeks
  Before starting the procedures, the participants were given verbal guidance on how to squeeze the dynamometers to ensure a maximum value. Then, the participants squeezed the dynamometer as hard as possible for three seconds. There were three measurements with 60-second pause intervals between the trials.
Total body fat (%) | 12 weeks
  Using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
Truncal body fat (%) | 12 weeks
  Using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
Muscle power | 12 weeks
  The peak power at 60°/s knee extension left, right (Nm/s), and flexion left, right (Nm/s) at baseline and after 12 weeks
Skeletal muscle mass (kg) | 12 weeks
  Using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
Short Physical Performance Battery total score | 12 weeks
  Short Physical Performance Battery total score at baseline and after 12 weeks. The Short Physical Performance Battery (SPPB) total score ranges from a minimum of 0 to a maximum of 12. A higher score indicates better physical performance, while lower scores reflect greater impairment in physical function. The SPPB assesses lower extremity function through balance tests, gait speed, and chair stand tests.
Gait speed (seconds) | 12 weeks
  Assessed by timing the participants as they walked 2.44 metres at their regular pace at baseline and after 12 weeks
Repeated chair stand test (seconds) | 12 weeks
  Timed as they completed five sit-to-stand repetitions at baseline and after 12 weeks
EuroQol five dimensional five levels | 12 weeks
  Index of life quality, minimum, maximum values (0, 1), higher scores mean a better outcome, which will be measured at baseline and after 12 weeks
Concentration of insulin-like growth factor 1 | 12 weeks
  Insulin-like growth factor 1 (ng/mL) measured at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea